CLINICAL TRIAL: NCT01557790
Title: A Phase II Study of Adjuvant Proton Radiation Therapy for the Treatment of Stage I, IIA and IIB Seminoma
Brief Title: Proton Radiotherapy for Stage I, IIA, and IIB Seminoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17811
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Stage I, IIA and IIB Seminoma
Keywords: Adult male; 18 years or older; clinical diagnosis
MeSH Terms: interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton RT (Experimental): Subjects receive proton radiation for seminoma
  Interventions: Radiation: Proton Radiation Therapy

INTERVENTIONS:
Radiation: Proton Radiation Therapy

SUMMARY:
Phase II study using Proton radiation therapy to treat males, aged 18 years or older, with Stage I, IIA and IIB Seminoma. This research study will be done in conjunction with the Robert H. Burr Proton Therapy Center at the Mass. General Hospital and the Department of Defense. In the feasibility portion of the study patients will be evaluated to determine acute toxicity. If the study is deemed feasible the principal investigator (PI) hopes that proton RT will reduce the lethargy rate as compared to photon radiation therapy (RT).

DETAILED DESCRIPTION:
This is a Phase II study using proton radiation therapy in addition to their standard care in subjects who have Stage I, IIA, IIB Seminoma. Testicular cancer are the most common solid cancers among men aged 20 to 35. Each subject must be 18 years of age or older and have a histologically proven diagnosis of testicular cancer. In addition to a subject's routine exams and tests, they will be asked to complete a series of quality of life questionnaires before, during and after their treatment. All side effects/toxicities will be monitored and recorded. Patients will be followed for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria

* Histological diagnosis; Histologically proven diagnosis of testicular seminoma; - Histologically confirmed seminomatous germ cell tumor of the testis categorized as either "classical" or "anaplastic;
* Stage I disease; Any pT N0 M0 S0-3 (Appendix B) [AJCC, 7th Ed.] (72); Stage IIA or IIB disease;
* Any pT N1 M0 S0-3 (Appendix B) [AJCC, 7th Ed.] (72); Any pT N2 M0 S0-3 (Appendix B) [AJCC, 7th Ed.] (72); (at the discretion of the principal investigators, bulky stage IIB may be excluded from the study, according to National Comprehensive Cancer Center Guidelines. 2. Laboratory evaluations; Semen analysis (patients will not be excluded if they do not wish to have an analysis or their insurance denies the claim) Follice-stimulating hormone (prior to the start of radiation) Luteinizing Hormone (Prior to the start of radiation) Lactate Dehydrogenase (Prior to the start of radiation) Human Chorionic Gonadotropic (Prior to the start of radiation) Complete blood count (Prior to the start of radiation) Testosterone (prior to the start of radiation) 3. Appropriate stage for protocol entry, as per protocol section 3.2.1, , based upon the following minimum diagnostic workup: History and physical examination, including a complete list of current medications; Chest x-ray (PA and lateral views) or CT Chest (within 3 months of study registration); Abdominal/pelvic CT scan or Abd/pelvic MRI(within 3 months of study registration); Brain MRI if clinically indicated; Bone scan if clinically indicated; 4. For stage I seminoma patients only, definitive surgical intervention within ten weeks prior to registration; Patients undergoing scrotal violations (scrotal orchiectomy, transscrotal biopsy, testicular fine needle aspiration, scrotal exploration) will be eligible; 5. The patient is a candidate for definitive external beam radiotherapy; The patient has had no prior radiotherapy to the region of study; The patient has no inflammatory bowel disease, active collagen vascular or connective tissue disorders, and no other medical or social contraindications to radiotherapy, as determined by a participating radiation oncologist; 6. Patient age: ³18 years; 7. Patient ECOG performance status: 0-1 (Appendix C); 8. For Stage II disease recurrence, rebiopsy is not clinically indicated. Imaging suffices for confirmation of recurrence

Exclusion Criteria

* Prior radiotherapy to the region of the study cancer
* Prior radiation therapy for a different cancer or disease process is allowed, provided there will be no overlap of radiation therapy fields between the participant's prior and current course of radiation therapy, radiotherapy was completed more than four weeks from first fraction of proton therapy administered in this study, and the participant has recovered to Grade ≤1 toxicity related to prior radiotherapy
* Chemotherapy administered for the diagnosis of seminoma
* Prior chemotherapy for a different cancer is allowed, provided therapy was completed more than twelve months from first fraction of proton therapy administered in this study and the participant has recovered to Grade ≤1 toxicity related to agents previously administered
* Incomplete definitive surgical orchiectomy, including diagnostic biopsy alone
* Pelvic lymph node dissection for the diagnosis of seminoma
* An investigational drug administered for the diagnosis of seminoma given concurrently or within four weeks of the first fraction of proton therapy administration
* Prior or concurrent second invasive malignancy other than non-melanoma skin cancer, unless disease free for a minimum of five years
* Known severe, active co-morbidity, defined as follows:Any clinically significant unrelated systemic illness, medical condition, or other factor, which at the discretion of the Principal Investigators, would interfere in the safe and timely completion of study procedures, compromise the patient's ability to tolerate the protocol therapy, or is likely to interfere with the study procedures or results
* Cognitively impaired patients who cannot provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Bekelman, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Jason Efstathiou, MD, Ph.D., Principal Investigator — Massachusettes General Hospital
Locations (2):
- United States (2):
  - Massachusettes General Hospital, Boston, Massachusetts
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton RT: Subjects receive proton radiation for seminoma
  Proton Radiation Therapy
Period: Overall Study
Arm/Group | Proton RT
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton RT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.86 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton RT
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Proton RT
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton RT (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Other Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (5)
Nausea (Gastrointestinal disorders) | 5 (8)
Work Stress (Social circumstances) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT01557790/Prot_SAP_000.pdf